CLINICAL TRIAL: NCT00420160
Title: Does Moderate Intensity Exercise Help Prevent Smoking Relapse Among Women?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Williams, Research Associate, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R03CA119747 (NIH)
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Lung Cancer; Heart Disease; COPD
Keywords: Smoking cessation; Exercise; Nicotine Patch; Disease Prevention
MeSH Terms: conditions — Lung Neoplasms; Heart Diseases; Pulmonary Disease, Chronic Obstructive; Smoking Cessation; Motor Activity

ARMS (2):
- Exercise (Experimental): 3x/wk 50 minutes of moderate intensity walking on treadmills + health education videos
  Interventions: Behavioral: Smoking cessation treatment plus moderate intensity exercise
- Health Education (Other): Contact control group attending 3x/wk 50 minutes of health education videos
  Interventions: Behavioral: Smoking cessation treatment plus health education

INTERVENTIONS:
Behavioral: Smoking cessation treatment plus moderate intensity exercise
  Arms: Exercise
Behavioral: Smoking cessation treatment plus health education
  Arms: Health Education

SUMMARY:
This study compares the effects of a standard smoking cessation treatment, including one-time brief counseling and provision of nicotine patch plus an 8-week moderate intensity exercise program versus the same standard smoking cessation treatment plus equivalent contact control among 60 healthy women. We hypothesize that participants in the smoking cessation plus moderate intensity exercise condition will be more likely to quit smoking than participants in the smoking cessation treament plus contact control condition.

DETAILED DESCRIPTION:
This study compares the effects of a standard smoking cessation treatment, including one-time brief counseling and provision of nicotine patch plus an 8-week moderate intensity exercise program versus the same standard smoking cessation treatment plus equivalent contact control among 60 healthy women. A number of techniques will be used to increase compliance with the treatment program, thus more effectively isolating the effects of exercise. These include: (1) a two-week run-in period prior to randomization; (2) use of behavioral contracting prior to participant randomization; and (3) performance of all exercise on-site. Smoking cessation outcomes (continuous abstinence and point prevalence abstinence) will be verified by carbon monoxide and saliva cotinine. Physical activity will be evaluated by attendance at the supervised sessions. We hypothesize that participants in the smoking cessation plus moderate intensity exercise condition will be more likely to quit smoking than participants in the smoking cessation treament plus contact control condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy sedentary smokers (> 4 per day for at least one year)
* Ages 18 to 65 years
* Must be able to give informed consent
* Must live in the area for the next 3 months
* Willing to use the nicotine patch to attempt smoking cessation
* Must receive consent to participate from primary care physician

Exclusion Criteria:

* Cannot read or write fluently in the English language
* Pregnancy or plans to attempt pregnancy
* 60 minutes or more per week of moderate or vigorous physical activity
* Smokes cigars, pipes, or uses smokeless tobacco at least once per week
* Currently in a quit smoking program
* Currently using NRT of any kind or using any other quit smoking method or treatment
* Never had an adverse reaction to the nicotine patch resulting in discontinuation of use
* Poor willingness or inability to comply with protocol requirements
* An employee of the Centers for Behavioral and Preventive Medicine
* Previous participant in Commit to Quit or Fit to Quit smoking cessation studies
* Another member of the household is or has been enrolled in this study
* Currently taking a medication that might impact heart rate response, including but not limited to:

Acebutolol Atenolol Carvedilol Metoprolol Nadolol Pindolol Propranolol Timolol

Medical problems:

* Cardiac disease of any kind such as angina, a history of myocardial infarction or valve disease including mitral valve prolapse. Anyone with an interventional procedure such as a stent
* Pain, discomfort (or other anginal equivalent) in the chest, neck, jaw, arms or other areas that may be due to ischemia
* Cerebrovasular disease such as stroke or history of transient ischemic attacks
* Peripheral vascular disease (such as claudication)
* Diabetes (both Type I and II)
* Chronic infectious disease (HIV, hepatitis) (hepatitis A is okay)
* Liver disease
* Cystic fibrosis (CF)
* Chronic obstructive pulmonary disease (COPD) (see asthma and bronchitis under questionable)
* Interstitial lung disease
* Emphysema
* Chronic Bronchitis
* Orthopnea (difficulty breathing except in the upright position) or paroxysmal nocturnal dyspnea (sudden shortness of breath at night typically triggered by lying down)
* Current diagnosis of Chronic Fatigue Syndrome
* Current diagnosis of Fibromyalgia
* Abnormal exercise stress test
* Hypertension (anyone currently being followed and/or treated for hypertension)
* Cancer treatment (other than skin cancer) within the past 6 months
* Musculoskeletal problems such as osteoarthritis, gout, osteoporosis or back, hip or knee pain that can interfere with physical activity (i.e., walking at a brisk pace - about 3-mph)
* Any other serious medical condition that might make exercise unsafe or unwise

Psychiatric Problems

* Hospitalization for a psychiatric disorder in the last 6 months
* Currently suicidal or psychotic, (or suicidal/psychotic in last 6 months)
* Self-report of more than three alcoholic drinks per day on 5 or more days; 5 or more alcoholic drinks on 3 or more days
* Taking these specific medications for psychiatric problems: Mood stabilizer (Lithium, Depakote, Neurontin), Antipsychotics (Haldol, Clozaril, Risperdal)
* Must be on other current psychiatric medications for at least three months

REQUIRES MD CONSENT FOR THE SPECIFIC CONDITION

* Lightheadedness, dizziness, vertigo, or fainting
* Last electrocardiogram (EKG) performed was abnormal
* Anemia
* Previous ETT for medical reason with normal results
* Irregular heart beats or palpitations in the past two years
* Heart murmurs in the past two years - the person will need physician's consent and an echocardiogram showing no evidence of significant heart disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence smoking abstinence verified by saliva cotinine taken | post-intervention (8 weeks after baseline)

SECONDARY OUTCOMES:
7-day point prevalence smoking abstinence verified by saliva cotinine | taken one month post-intervention (12 weeks after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: David M Williams, Ph.D., Principal Investigator — The Miriam Hospital and Brown Medical School
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Williams DM, Whiteley JA, Dunsiger S, Jennings EG, Albrecht AE, Ussher MH, Ciccolo JT, Parisi AF, Marcus BH. Moderate intensity exercise as an adjunct to standard smoking cessation treatment for women: a pilot study. Psychol Addict Behav. 2010 Jun;24(2):349-54. doi: 10.1037/a0018332. PMID 20565161
- [Result] Williams DM, Dunsiger S, Whiteley JA, Ussher MH, Ciccolo JT, Jennings EG. Acute effects of moderate intensity aerobic exercise on affective withdrawal symptoms and cravings among women smokers. Addict Behav. 2011 Aug;36(8):894-7. doi: 10.1016/j.addbeh.2011.04.001. Epub 2011 Apr 15. PMID 21543158